CLINICAL TRIAL: NCT06554093
Title: A Prospective, Dual Canter, Double Armed, Open Label, Clinical Study to Evaluate the Performance of the PathKeeper System for Pedicle Screw Positioning in Spine Surgery
Brief Title: Study Comparing the PathKeeper System for Pedicle Screw Positioning in Spine Surgery With Traditional Care
Acronym: PKSforPSP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deep Health Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL0003; 341268 (Other: IRAS(Integrated research application system))
Record Dates: First submitted 2024-03-12; First posted 2024-08-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-08

CONDITIONS: Scoliosis; Scoliosis; Adolescence; Scoliosis Kyphosis; Scoliosis Lumbar Region; Scoliosis Thoracic Region; Pathologic Fracture
Keywords: fusion; screw positioning; screw insertion
MeSH Terms: conditions — Scoliosis; Fractures, Spontaneous

STUDY DESIGN:
Intervention Model Description: • Experimental arm: PathKeeper System (PKS) One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under PKS intraoperative navigation guidance.
  Intervention: Medical Device - PKS. The PKS spine navigation system is for spatial positioning and orientation of surgical instruments during pedicle screw instrumentation in patients undergoing posterior fusion in single or multiple levels.
  • Control arm: Standard of care - free-hand technique guided by intra-operative 2D Fluoroscopy One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under free-hand technique guided by intra-operative 2D fluoroscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Device- PathKeeper System (PKS) (Experimental): One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under PKS intraoperative navigation guidance.
  Intervention: Medical Device - PKS. The PKS spine navigation system is for spatial positioning and orientation of surgical instruments during pedicle screw instrumentation in patients undergoing posterior fusion in single or multiple levels.
  Interventions: Device: Medical Device - PKS
- 2D Fluoroscopy (Active Comparator): Control arm: Standard of care - free-hand technique guided by intra-operative 2D Fluoroscopy One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under free-hand technique guided by intra-operative 2D fluoroscopy
  Interventions: Device: Medical Device - PKS

INTERVENTIONS:
Device: Medical Device - PKS — The PKS spine navigation system is for spatial positioning and orientation of surgical instruments during pedicle screw instrumentation in patients undergoing posterior fusion in single or multiple levels.
  Other Names: Device- Fluoroscopy

SUMMARY:
The goal of this is to evaluate performance of the Pathkeeper Surgical System. The main question[s]it aims to answer are: 1) evaluate pedicle screw position Participants will in compare Experimental arm: PathKeeper System (PKS) with control arm

DETAILED DESCRIPTION:
Trial design

* Allocation: Randomized
* Interventional Model: Parallel Assignment (double armed)
* Interventional Model Description: Dual center, prospective, randomized cohort study.
* Masking: None (Open Label)
* Primary Purpose: Treatment
* Enrolment: 32 (thirty-two) patients - 16 (sixteen) patients experimental and 16 control arms (100 screws each arm, estimated 20% of patients drop out).

Study arms

1. Experimental arm: PathKeeper System (PKS) One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under PKS intraoperative navigation guidance.

   Interventions: Medical Devise - PKS. The PKS spine navigation system is for spatial positioning and orientation of surgical instruments during pedicle screw implantation in patients undergoing posterior fixation in single or multiple levels.
2. Control arm: free-hand technique guided by intra-operative 2D Fluoroscopy One to ten-level posterior, open, instrumented spine surgery using unilateral or bilateral pedicle screw instrumentation under free-hand technique guided by intra-operative 2D fluoroscopy.

Interventions: Pedicle screws will be placed using the free-hand technique with 2D fluoroscopy as the intraoperative imaging modality.

Primary endpoints:

Evaluate and classify the pedicle screw positions as per the Gertzbein-Robbins classification scale based on a low-dose post-operative CT scan, in each study arm and comparatively.

Number of misaligned screws as per the Gertzbein-Robbins classification scale (Gertzbein and Robbins, 1990) class E screws class D screws class C screws class B screws class A screws

Secondary endpoints:

1. Evaluate radiation exposure dose and time in the operating room during the procedure in each study arm and comparatively.
2. Evaluate time-per-screw for the experimental device arm (PKS) arm.
3. Length of stay - (non-critical)
4. Estimated blood loss (EBL) - (non-critical)
5. Number of reported complications (neurological deficits, dural tears, deep wound infections, etc.) while hospitalized

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 16 and above years old
* Patients who are about to undergo open, instrumented spinal surgery
* Signed informed consent form

Exclusion Criteria:

* Men and women
* 16 and above years old
* Patients who are about to undergo open, instrumented spinal surgery
* Signed informed consent form

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the screw implantation by Gertzbein-Robbins scale | Post-operative CT scan to be performed before hospital discharge and evaluation can be done right after or at the end of the of the data collection
  Mean and STD of Gertzbein-Robbins classification scale based on a low-dose post-operative CT scan

SECONDARY OUTCOMES:
Evaluate radiation exposure dose and time in the operating room during the procedure in each study arm and comparatively. | 24 hours after surgery
  Mean and STD Values in milli-gray (mGy) and seconds collected from the c-Arm
Evaluate time-per-screw for the experimental device arm (PKS) arm. | Values to be collected during each surgery once the last screw insertion is completed (1-2 hours within the surgery)
  Operative time per screw

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To be done